CLINICAL TRIAL: NCT01544660
Title: Bone Quality by vQCT and HR-pQCT:Translation to Multi-center Clinical Research
Acronym: Interscanner
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: NIH-Multicenter Interscanner
Record Dates: First submitted 2012-02-14; First posted 2012-03-06 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Bone Mineral Density
Keywords: spine and hip scan; BMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Scanning: no treatment
- scanning: no treatment

SUMMARY:
Our overarching aim is to set up a procedural, analytic and developmental framework to establish CT of the central and peripheral skeleton as a clinically useful biomarker for skeletal strength in the clinical research and ultimately in the clinical setting. To accomplish this, the investigators will develop and validate phantoms and scanning procedures to standardize strength and structure measurements between different vQCT scanners and develop standardized acquisition, analytical, and quality control techniques for HR-pQCT with an emphasis on optimization for multi-center studies.

DETAILED DESCRIPTION:
The investigators will develop new calibration phantoms to address inter and intra scanner variability in vQCT and HRpQCT. Phantom sets to evaluate inter-scanner disparity and determine corrections to apply to in vivo scan data in the multi-center settings. These methods will be validated in a multi-center phantom study and in a 120 patients

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* must be able to lie down on bed

Exclusion Criteria:

* on wheel chair
* age above 80 years 0r less than 65 years

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy men and women aged 65-80
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Develop and Validate phantoms and scanning procedures to standardize strength and structure measurements between different scanners. | one visit lasting 3 hours for each subject.
  Correction of the in vivo images using the proposed inter-scanner calibration approaches will improve the quality of multi-site data by reducing the variability in CT structure and strength measures. To study the Multi-center standardization of vQCT and HR-pQCT imaging we will develop new calibration phantoms to address inter and intra-scanner variability in vQCT and HRpQCT bone strength and structure estimates.

SECONDARY OUTCOMES:
Development of open-source image analysis metric for vQCT | Time frame will be 3 hours for a visit
  To provide standardized analysis of future clinical studies and retrospective analysis of past trials, we will develop a set of image analysis metrics for vQCT (trabecular, cortical and integral BMD, cortical thickness, cross-sectional areas, axial and bending strength estimates). These metrics will be made available to the community in an open source format, allowing them to be incorporated into commercial software platforms at the discretion of the manufacturer, incorporation as a plug-in for NIH supported programs such as MIPAV.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lang, Principal Investigator — University of California, San Francisco
Locations (1):
- Department of Radiology, UCSF, San Francisco, California, United States